CLINICAL TRIAL: NCT02556398
Title: Use of Mobile-based Technologies to Improve Diabetes Self-management and Postprandial Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-07
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention - Educ Module and App (Experimental): Participants in this arm to be given smartphone app ("Sugar Sleuth") and educational module.
  Interventions: Behavioral: Sugar Sleuth

INTERVENTIONS:
Behavioral: Sugar Sleuth — Educational module and use of smart phone app ("Sugar Sleuth")

SUMMARY:
The project involve evaluation of a web-based nutrition education program and pilot-testing of a new smartphone app for real-time data logging to identify factors causing glycemic variability.

DETAILED DESCRIPTION:
The intervention will be three (3) months in duration and will entail use of a smart phone app for real-time data logging to identify factors causing glycemic variability, as well as use of a web-based nutrition education program. The investigators postulate that the interactive nutrition education curriculum - which will provide feedback to patients about the inter-relationship between their food intake and postprandial glucose profiles, as well as practical guidance for improvements - will lead to a change in food choices and improved post-prandial glucose control.

ELIGIBILITY:
Inclusion Criteria

Individuals that satisfy all of the following conditions will be considered for participation:

1. Must be between the ages of 25 - 75 years of age (inclusive)
2. Type 1 diabetes diagnosis at least 1 year, treated with multiple daily injections or insulin pump.
3. A1c 7.5-9.0%

Exclusion Criteria

1. Current or past use of real-time CGM for more than 2 months.
2. Pregnancy (self-reported) or planning conception in next 6 months.
3. History of disordered eating, actively trying to lose weight or planning to do so, BMI > 30 kg/m2 (to limit participation by individuals who are actively trying to lose weight),
4. Medical conditions or medications that would affect gastric emptying such as gastroparesis, bariatric surgery, medications such as pramlinitide, liraglutide or exenatide.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) above target (> 180 mg/dL) | 3 months
  Amount of time spent above >180 mg/dL on CGM Freestyle Libre readings

CONTACTS AND LOCATIONS:
Overall Officials: Elena Toschi, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT02556398/ICF_000.pdf